CLINICAL TRIAL: NCT04609371
Title: Assisting Family Physicians With Gaps in Mental Health Care Generated by the COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: PanDirect: Self-care Tools and Telephone Coaching for Depression and Anxiety During Pandemics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Responsible Party: Principal Investigator, Mark Yaffe, Professor, Department of Family Medicine, McGill University and Family physician, St. Mary's Hospital Center, St. Mary's Research Center, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMHC-20-10
Record Dates: First submitted 2020-10-19; First posted 2020-10-30 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Mental Health Wellness 1; Coaching; Pandemic; Depression, Anxiety; Self-care Tools
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-care tools (Experimental): Arms Assigned Interventions Experimental: self-care tools
  The tools are adapted from those successfully deployed in the DIRECTsc depression self-care project focusing on patients with depressive symptoms, but abbreviated to meet the needs of the proposed short-term intervention for a broader sample of patients to include those with anxiety symptoms and with minimal symptoms. Tools will include individual chapters of the Antidepressant Skills Workbook; the mood monitoring tool; a workbook on managing worry; relaxation audio files and information on exercise and healthy eating. In view of the short duration of the intervention (8 weeks), a maximum of 2 tools will be sent to each participant.
  An algorithm will determine which self-care tools, matched to the specific mental health symptoms reported by participants, will be sent to the participants.
  Interventions: Behavioral: self-care tools
- coaching (Experimental): Participants will receive the algorithm-determined self-care tools, matched to the specific mental health symptoms reported by participants as in the first arm. They will ALSO be offered up to 3 coach calls. Coaching by a trained lay coach will be structured and guided by a manual. Trained lay coaches will call participants in the week following delivery of the toolkit to guide them through the self-care toolkit over an 8-week period. Coaches will contact participants a maximum of 3 times, with calls expected to average 15-20 minutes. Call content will be guided by a structured coaching manual adapted from those used in the team's previous two RCTs of the self-care materials. The coaches will follow structured agendas, keep records of all contacts.
  Interventions: Behavioral: self-care tools; Behavioral: lay telephone coaching

INTERVENTIONS:
Behavioral: self-care tools — self-care tools only
Behavioral: lay telephone coaching — coaching
  Arms: coaching

SUMMARY:
During pandemics older adults with chronic physical conditions are a particularly vulnerable population for unmet mental health needs. This is a consequence of a number of factors which include decreased access to their doctors because of restrictions in visits in order to decrease risk of disease transmission and because doctors are seconded to provide medical services in areas of high priority. Since Public Health authorities worry that pandemics may be a reality of the future, this study is being operationalized during the present COVID-19 pandemic in order to see what can be learned about different ways to provide mental health care under such constraints.

The study offers evidence-based approaches to managing feelings of anxiety or depression that may have existed prior to the onset of a pandemic, or that have arisen during a pandemic. It uses principles of cognitive behavioural therapy in which participants are offered self-care tools to help them develop strategies for dealing with their various symptoms. These tools have already been shown by the team to be effective in other contexts in studies DIRECT-sc (Effectiveness of a supported self-care intervention for depression compared to an unsupported intervention in older adults with chronic physical illnesses) and CanDIRECT (Effectiveness of a telephone-supported depression self-care intervention for cancer survivors).

The present study, PanDIRECT (Assisting Family Physicians with Gaps in Mental Health Care Generated by the COVID-19 Pandemic), aims to answer the following questions:

1. Can these tools be used in the community care of mental health problems during pandemics?
2. Are they acceptable to patients?
3. Using a randomized control trial, does lay-coaching of use of these tools improve their use and patient outcomes?
4. Do family practitioners value patient information sent to them at the end of the trial

ELIGIBILITY:
Inclusion Criteria:

* 65+ years old
* consented to be recontacted (participant in a previous study)

Exclusion criteria:

* moderate to severe cognitive impairment (using BOMC a brief cognitive screen) -unable to read in English or French (self-reported); hearing impairment (as judged by research staff);
* currently receiving counseling or psychological therapy (as these treatments may conflict with the self-care interventions)
* currently living in a long term care or other medicalized facility,
* presenting suicidal intent (as identified through the final item of the PHQ-9 which will be asked at screening).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Consent rate | At recruitment
  Number of consenting participants out of total number contacted over the recruitment period
Data completion rate | From recruitment launch to completion of follow-up (4 months)
  Investigators will report on rates of missing data from baseline and follow-up questionnaires
Fidelity of intervention completion | A 8 week follow-up
  Logs and checklists will be used to evaluate completion of intervention, as per protocol
Severity of depression symptoms | At baseline
  Using the validated 9 item Patient Health Questionnaire (PHQ-9). Scores range from 0 to 27 - higher score indicates more severe depression
Severity of depression symptoms | At 8 week follow-up
  Using the validated 9 item Patient Health Questionnaire (PHQ-9). Scores range from 0 to 27 - higher score indicates more severe depression
Severity of anxiety symptoms | At baseline
  Using the validated 7 item General Anxiety Disorder (GAD-7) instrument. Scores range from 0 to 21 - higher score indicates more severe anxiety
Severity of anxiety symptoms | At 8 week follow-up
  Using the validated 7 item General Anxiety Disorder (GAD-7) instrument. Scores range from 0 to 21 - higher score indicates more severe anxiety
Use of health care services | At baseline
  Using questions developed by the team and administrative databases to assess use of hospital and mental health care services
Use of health care services | At 8 week follow-up
  Using questions developed by the team and administrative databases to assess use of hospital and mental health care services
Use of the self-care materials | At 8 week follow-up
  Using adherence questions developed by the team, not scored

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's Hospital Research Centre, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No